CLINICAL TRIAL: NCT04996914
Title: Adjuvant Stereotactic Body Radiation Therapy After Trans-arterial Chemoembolization in Hepatocellular Carcinoma
Acronym: ASTrH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-341
Record Dates: First submitted 2021-07-02; First posted 2021-08-09 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma Non-resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE+SBRT. (Experimental): If a patient is eligible to participate in the project according to the in- and exclusion criteria, the patient will assigned to 1-2 sessions of TACE followed by SBRT within one month from last TACE session .
  Interventions: Procedure: TACE; Radiation: SBRT

INTERVENTIONS:
Procedure: TACE — 1-2 session TACE before SBRT according to the preference of the interventional radiologist. Goal of TACE is the complete emnbolization of the HCC-nodules. It is allowed to use both conventional TACE (cTACE) and drug-eluting beads TACE (DEB-TACE) according to the interventional radiologist preference.
Radiation: SBRT — SBRT should be 1 month after last TACE. This can be extended till 2 months if indicated. However, prolongation of the gap between TACE and SBRT is not encouraged.
  Treatment center should choose one of fractionation schedule mentioned allowed in the study, in order to achieve a balance between dose applied for tumor control and constraints for OAR PTV Dose in 5 / 8 fractions (Gy) EQD2 (α/β 10Gy) 5x 8-6 Gy @ 83% isodose = 40-30 Gy (60-40 Gy) 8 x 6-4.5 Gy @ 83% isodose = 48-36 Gy (64-43.5 Gy)

SUMMARY:
The study investigates the adjuvant SBRT following TACE in early and intermediate stages HCC not amenable for surgical resection or orthotopic liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* HCC (diagnosis: histological or radiological)
* Age: 18-80
* Number of lesions 1-3 lesions
* Size of the lesion (or sum of 2-3 lesions) ≥ 4 cm
* Sufficient non-tumorous liver volume (≥ 800 cm3)
* Child Pugh Score: A5-6 or B7-8
* BCLC A or B
* Patient is illegible or refused surgical resection or orthotopic liver transplant
* Blood work (within 2 weeks before registration):
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm³)
* Platelets ≥50,000 cells/mm³
* AST (and ALT) < 5 times ULN
* Serum creatinine ≤ ULN or creatinine clearance ≥ 50 mL/min

Exclusion Criteria:

* Evidence of extrahepatic disease (lymph node or distant metastases)
* Evidence of macroscopic vascular invasion
* Evidence of an arterio-portal or arterio-venous fistulas
* History of previous malignancy
* Previous SIRT
* Previous Sorafenib in the last 8 weeks
* Pregnant and lactating females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
1-year local control rate | 12 Months
  After one year from the treatment, the precentage with alive subjects with no signs of local progression (the irradiated lesion).
  Local progression defined as more than 20% increase in diameter of enhancing tumor on contrast-enhanced CT scan in arterial phase or a new tumor mass within the original tumor volume according to modified RECIST criteria (mRECIST)

SECONDARY OUTCOMES:
Qualtiy of life based on EORTC QLQC30 | 12 Months
  alive subjects will fill quality of life questionnaires (EORTC QLQC30) before the treatment and after 3,6 and 12 months after.
  The results before and after the treatment will be presented in comaprsion to the reference data.
1- year progression free survival | 12 Months
  After one year from the end of the treatment, the percentage of alive subjects without the apperance of new hepatic and/or extra-heaptic new lesions outside the SBRT-field.
  This will be measured using contrast-enhanced CT scan Liver/Abdomen and Thorax
Quality of life based on EORTC QLQ-HCC18 | 12 Months
  alive subjects will fill quality of life questionnaires (EORTC QLQ-HCC18) before the treatment and after 3,6 and 12 months after.
  The results before and after the treatment will be presented in comaprsion to the reference data.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Eble, Professor Dr. med., Study Chair — University medical center RWTH Aachen; Philipp Bruners, Professor Dr. med., Study Chair — University medical center RWTH Aachen; Ahmed Allam Mohamed, MBBS, MSc, MD, Study Chair — University medical center RWTH Aachen; Oliver Beetz, Prof. Dr.med . MHBA, Study Chair — University medical center RWTH Aachen; Marie-Luise Berres, Prof. Dr.med., Study Chair — University medical center RWTH Aachen

IPD SHARING:
Plan to Share IPD: Undecided